CLINICAL TRIAL: NCT06265090
Title: Effect of Lumbar Stabilization Exercises Combined With Ball and Balloon Exercise in Treatment of Chronic Non-specific Low Back Pain: Randomized Clinical Trial
Brief Title: Effect of Lumbar Stabilization Exercises Combined With Ball and Balloon Exercise in Treatment of Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F.P.T 2307017
Record Dates: First submitted 2024-01-17; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-01

CONDITIONS: Chronic Mechanical Low Back Pain
MeSH Terms: interventions — Exercise Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: This randomized controlled experimental trial was carried out at the outpatient clinic of faculty of physical therapy, Delta University for science and technology from April 2023 to October 2023. The aims of the study and the study protocol were explained for each patient before participation in the study. All patients signed an approved informed consent form for participation in this study. Before starting the treatment program, a complete history and physical examination will be taken for all patients.
  Subjects:
  Seventy male and female physiotherapy students have chronic non-specific low back pain will be chosen from faculty of physical therapy, delta university for science and technology.
  The local ethics committee approved this study (Delta University for science and technology, faculty of Physical Therapy, Ethics committee F.P.T 2307017).
Who Masked: Participant, Care Provider, Investigator
Masking Description: the participants were selected randomly without their knowledge about in experimental or control group the assessor was for assessment only and the therapist was for treatment only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ball and balloon exercises (Experimental): Ball and balloon exercise exercises:
  The second group received hemibridge with ball and balloon exercise in combination to core stability exercises.
  Instructions
  1. supine-lying position, feet up against a wall, and bend your knees as well as hips to a 90° angle.
  2. Insert a ball measuring between four and six inches in diameter in the space between your knees.
  3. Put your left hand upon a balloon and your right arm above your head.
  4. Tilt your pelvis to make sure your tailbone is just slightly elevated off the ground while you inhale with your nose and exhale using your mouth. Keep your low back as flat as possible on the mat. Dig your heels into the wall instead of pushing your feet flat.
  5. drop your left knee till it is below the level of your right, without moving your feet. the activation of your left inner thigh muscle.
  Interventions: Other: therapeutic exercises; Other: exercises
- core stability exercises (Active Comparator): Core stability exercises (CSE): Subjects in this group were handled with core stability exercises that targeted deep abdominal muscles. This included a series of exercises as well as a baseline therapeutic management of ultrasonic as well as TENS. A physiotherapist supervised these exercises.
  For four weeks, all groups did core stability exercises for 30 minutes three times per week.exercises. Based on the patient's success, the intensity of the individual training steadily increased with decreasing therapist support. Patients were told to contract their abdominal muscles and hold the contraction while continuing to breathe normally during each repetition of each exercise.
  Interventions: Other: therapeutic exercises; Other: exercises

INTERVENTIONS:
Other: therapeutic exercises — Protocol of hemibridge with ball and balloon exercise Participants were given exercise called as hemibridge with ball and balloon exercise for 3 sessions over 3 days/week.
  Other Names: core stability exercises
Other: exercises — The second group received hemibridge with ball and balloon exercise in combination to core stability exercises.
  Protocol of hemibridge with ball and balloon exercise The hemibridge with ball as well as balloon exercise was provided to the participants over the course of three sessions per week.
  Instructions
  1. supine-lying position, feet up against a wall, and bend your knees as well as hips to a 90° angle.
  2. Insert a ball measuring between four and six inches in diameter in the space between your knees.
  3. Put your left hand upon a balloon and your right arm above your head.
  4. Tilt your pelvis to make sure your tailbone is just slightly elevated off the ground while you inhale with your nose and exhale using your mouth. Keep your low back as flat as possible on the mat. Dig your heels into the wall instead of pushing your feet flat.
  5. drop your left knee till it is below the level of your right, without moving your feet. the activation of your left inner thigh muscle.
  Other Names: ball and balloon exercises

SUMMARY:
[Background] Low back pain occurs when a poor lifestyle weakens the muscular strength of the waist and excessive loads on and tensions of the muscles create pain. Mediating muscle weakening to stabilize the trunk is an important aspect in the recovery of body function in patients with LBP [Purpose], this study was conducted to investigate the effect of core stability exercises combined with ball and balloon exercises on chronic non-specific low back pain. [Subjects and Methods] a sixty patient of chronic non-specific low back pain were randomly assigned into two groups, group (A) received core stability exercises combined with ball and balloon exercises and group (B) received core stability exercises, these exercises were performed for three times a week for four weeks. Pain was assessed by visual analogue scale (VAS). Spinal function was measured by Arabic Oswestery Disability Index (AODI) and pulmonary function was assessed by pulmonary function test including forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), FEV1/FVC, maximum voluntary ventilation (MVV) and peak expiratory flow (PEF) before and after the study.

Keywords: core stability exercises, ball and balloon exercises, chronic non-specific low back pain

DETAILED DESCRIPTION:
Low back pain (LBP) is a common musculoskeletal disorder, with a current incidence of 60-90%; more than 80% of people will suffer LBP at some point in their lives. Approximately 15% of them suffer from chronic LBP. LBP arises when a poor lifestyle reduces the muscular power of the waist and causes discomfort from too much stress on and tensions in the muscles. Mediating muscular weakness to support the trunk is a key part of LBP patients' recovery of bodily function.

The most frequent type of low back pain has no clear cause. It is a type of pain in which imaging studies do not provide any useful information for treatment and are incapable of determining an accurate patho-anatomical diagnosis.

Supervised exercise therapy is recommended as a first-line treatment in the European recommendations and other clinical practice recommendations for the management of chronic non-specific low back pain (NSLBP). In order to restore appropriate kinetic function, core stability exercises have gained popularity as a type of therapeutic exercise. Core stabilization exercise is more effective than routine physical therapy exercise in terms of greater reduction in pain in patients with non-specific low back pain. Spinal stability is obtained from trunk muscular activity, and active simultaneous contractions are essential to promote spinal stability in low back pain patients with unstable lumbar regions. Excessive stress or higher mobility of the joints is generated by less movement of the vertebral joints; additionally, if the muscles that surround the vertebral column are unable to effectively manage this increased mobility, risk can arise. This epidemiological process can emerge in diverse forms in all vertebral joints and has a significant impact on spinal column functional alterations. Patients with back pain who sit for lengthy periods of time or have bad posture are more likely to develop kyphosis of the back joints and impaired flexibility.

A cross-sectional study was undertaken to assess changes in breathing, respiratory strength and endurance, core stability, diaphragm mobility, and chest expansion in NSLBP patients, and it was found that there was a significant link between impaired respiratory function and NSLBP.

The respiratory muscles, internal oblique, abdominal muscles, back fibers, and spinal multifidus are among the trunk muscles that help to support the spine. The pelvic floor muscles influence spinal stability by collaborating with the trunk muscles to generate abdominal pressure. The transversus abdominis muscle moves up and down while breathing and is the most important muscle required for preventing inspiration among the various muscles that contribute to spinal stability.

The relationship between respiratory muscles and trunk stabilization creates intra-abdominal pressure, which influences waist stability and safeguards the trunk muscles. Additionally, the pelvic floor muscles will contract if intra-abdominal pressure rises as a result of breathing exercises that stimulate the diaphragm. Therefore, even the deep stabilizing muscles can be easily activated when the abdominal muscles contract during breathing.

Materials and Methods

This randomized controlled experimental trial was carried out at the outpatient clinic of faculty of physical therapy, Delta University for science and technology from April 2023 to October 2023. The aims of the study and the study protocol were explained for each patient before participation in the study. All patients signed an approved informed consent form for participation in this study. Before starting the treatment program, a complete history and physical examination will be taken for all patients.

Subjects:

Seventy male and female physiotherapy students have chronic non-specific low back pain will be chosen from faculty of physical therapy, delta university for science and technology.

Inclusion criteria: 1- both male and female physiotherapy students of age from 18 to 25 years, 2- patients with low back pain with or without referred leg pain, 3- patients with low back pain more than 6 months.

Exclusion criteria: 1- patients with acute low back pain, 2- patients with lumbar disc prolapse, 3- patients with systemic disease or T.B 4- history with spinal fractures or spinal surgeries, 5- patients with spondylolithesis, 6- patients with sacroiliac dysfunction, 7- osteoporotic patients, 8- patients with spinal deformities, 9- patients had previously received physical therapy treatment for low back pain in a period of six months, 10- patients with pulmonary diseases.

The local ethics committee approved this study (Delta University for science and technology, faculty of Physical Therapy, Ethics committee F.P.T 2307017).

Sample size:

Arabic Oswestery Disability Index (AODI) was considered as the primary outcome in this study and used for calculating the sample size (using the G*power program 3.1.0 for two tails, paired test). The estimated sample (power of 60% and a significant alpha level of 95%) required a total of 60 participants. Therefore, at least 30 participants with NS-LBP were required for an each group. However, 10 patients were added to the sample size to account for the possibility of drop-outs. Therefore at least 35 participants per group were examined. Patients were randomly assigned into two groups through computer software. We put 70 patients on the software program and the program assigned it randomly. The first group (group A) was treated by core stability exercises in addition to physical therapy interventions. Second group (group B) was treated by core stability exercises combined with ball and balloon exercises in addition to physical therapy interventions, which will be only given 3 times/week for 4 consecutive weeks.

Assessment instrumentation:

Arabic Oswestery Disability Index (AODI) for functional assessment , visual analogue scale for pain and pulmonary function test

AODI assessment: Patients filled out a questionnaire that provides a percentage score of how well they functioned in everyday activities before and after sessions. This survey evaluates daily function in ten activities of daily living. The categories were scored from zero to five (6 categories). If all 10 sectors were finished the result is calculated as follows: if 20 the total result out of 50 total possible score x 100 = 40%.

Scores: 1- Zero to twenty percent: Minimal disability. 2- Twenty one to forty percent: Moderate disability. 3- Forty one to sixty percent: Severe disability. 4- Sixty one to eighty percent: Crippled 5- Eighty one to one

Visual Analogue Scale: The Visual Analogue Scale (VAS), a reliable and effective measure of pain intensity that is sensitive to variations in pain caused by clinical conditions, was used to assess the severity of the pain. At the scale's left end, a zero means there is no pain, and a 10 means the most agonizing suffering possible. A minor improvement with a change of 1.1-1.2 cm is clinically meaningful.

Pulmonary function tests: investigators used a Spirometry Medisoft ergocart professional, power 230V AC 50Hz, Serial number: 161121-05-0018, Belgium to assess pulmonary function, including forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), FEV1/FVC, maximum voluntary ventilation (MVV) and peak expiratory flow (PEF). The patients were taught the following procedure of doing PFT: (1) In order to prepare the patient, it was necessary to describe the test's goal and procedure in straightforward language and in a concise manner. (2) A clean mouthpiece was given to the patient and is attached to the valve at the end of the spirometer tubing.. (3) The patient was wearing a nasal clip, sitting comfortably with his or her feet flat on the ground; (4) The proper chin neck posture was demonstrated to the patient: the chin should be lifted and the neck slightly extended, and this position should be maintained during the forced expiratory procedures; the patient should not lean the chin to the chest. (5) The mouthpiece was inserted into the patient's mouth, but the patient was instructed not to bite down on it. The lips were also instructed to be tightly sealed, and the tongue was not to protrude into the mouthpiece. (6) The patient was instructed to inhale completely (must be completely full), followed by a quick and forceful exhalation through the mouthpiece. (7) It was recommended to perform at least three technically sound maneuvers, ideally with less than 0.15-L variation in FEV1 (and FVC) between the best and second-best result (get the best of 3). Each test was considered valid if it satisfies the repeatability and acceptability requirements listed below. The ventilatory reserve was measured by MVV, The patient was instructed on how to measure MVV by repeating steps 1 through 5 and then being instructed to breathe as quickly as forcefully as they can for 10-15 seconds.

Intervention Core stability exercises (CSE): participants in this group were handled with core stability exercises that targeted deep abdominal muscles. This included a series of exercises as well as a baseline therapeutic treatment of ultrasound and TENS. A physiotherapist supervised these exercises.

For four weeks, all groups did core stability exercises for 30 minutes three times per week. Isometric contraction was sustained for 7-8 seconds for each exercise. Each exercise was repeated ten times, with a three-second rest break between repetitions. Patients were given a 1-minute break between exercises.(20) Based on the patient's success, the intensity of the individual training steadily increased with decreasing therapist support. Patients were told to tense their abdominal muscles and hold them while continuing to breathe normally during each repetition of each exercise. All exercise sessions were performed in individual exercise programs with the therapist, and recorded in a diary to facilitate adherence rates. Abdominal hollowing, Side Bridge, supine extension bridge, straight leg rise from prone, alternate arm and leg raise from quadruped, and prone bridge were the core stability exercises. The CSE approaches are presented in Table 1.

Ball and balloon exercise exercises:

The second group received hemibridge with ball and balloon exercise in combination to core stability exercises.

Protocol of hemibridge with ball and balloon exercise Participants were given exercise called as hemibridge with ball and balloon exercise for 3 sessions over 3 days/week.

Instructions

1. Lie on your back with your feet against a wall and your knees and hips bent at a 90° angle.
2. Place a 4-6" ball between knees
3. Place your right arm over your head and a balloon in your left hand.
4. Inhale through your nose and exhale through your mouth, tilting your pelvis so that your tailbone is raised slightly off the surface. Maintain a flat low back on the mat. Instead of pressing your feet flat against the wall, dig down with your heels.
5. Shift left knee down so that it is below the level of right without moving feet. should feel left inner thigh engage.
6. Take right foot off the fall with left knee bent and you should feel the back of the left thigh engage. For the duration of the exercise, hold this posture.
7. Now breathe in through your nose and release softly into the balloon.
8. Hold your tongue on your roof of mouth for three seconds to stop the balloon from losing air.
9. Inhale once again via your nose without pinching the balloon's neck and while maintaining your tongue resting on the roof of your mouth.
10. Slowly blow out while fixing the balloon with hand.
11. Avoid using your cheeks or neck as a strike.
12. Pinch the balloon neck and take it out of your mouth after the fourth breath. Release the balloon's air.
13. Unwind and do the sequence four more times.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female physiotherapy students of age from 18 to 25 years
* Patients with low back pain with or without referred leg pain
* Patients with low back pain more than 6 months.

Exclusion Criteria:

* patients with acute low back pain
* patients with lumbar disc prolapse
* patients with systemic disease or T.B 4- history with spinal fractures or spinal surgeries,
* patients with spondylolithesis,
* patients with sacroiliac dysfunction,
* osteoporotic patients
* patients with spinal deformities
* patients had previously received physical therapy treatment for low back pain in a period of six months
* patients with pulmonary diseases.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
visual analogue score | pre the intervention and immediately after the intervention
  The Visual Analogue Scale (VAS), a reliable and effective measure of pain intensity that is sensitive to variations in pain caused by clinical conditions, was used to assess the severity of the pain. At the scale's left end, a zero means there is no pain, and a 10 means the most agonizing suffering possible. A minor improvement with a change of 1.1-1.2 cm is clinically meaningful.

SECONDARY OUTCOMES:
forced expiratory volume in the first second (FEV1) in liters | pre the intervention and immediately after the intervention
  Pulmonary function tests: We used a Spirometry Medisoft ergocart professional, power 230V AC 50Hz, Serial number: 161121-05-0018, Belgium to assess pulmonary function, including forced expiratory volume in the first second (FEV1) The patients were taught the following procedure of doing Pulmonary Function Test: (1) A clean mouthpiece was given to the patient and is attached to the valve at the end of the spirometer tubing.. (2) The patient was wearing a nasal clip, sitting comfortably with his or her feet flat on the ground; (3) The proper chin neck posture was demonstrated to the patient: the chin should be lifted and the neck slightly extended, and this position should be maintained during the forced expiratory procedures
forced vital capacity (FVC) in liters | pre the intervention and immediately after the intervention
  Pulmonary function tests: We used a Spirometry Medisoft ergocart professional, power 230V AC 50Hz, Serial number: 161121-05-0018, Belgium to assess pulmonary function, includingforced vital capacity (FVC) The patients were taught the following procedure of doing Pulmonary Function Test: (1) In order to prepare the patient, it was necessary to describe the test's goal and procedure in straightforward language and in a concise manner. (2) A clean mouthpiece was given to the patient and is attached to the valve at the end of the spirometer tubing.. (3) The patient was wearing a nasal clip, sitting comfortably with his or her feet flat on the ground; (4) The proper chin neck posture was demonstrated to the patient: the chin should be lifted and the neck slightly extended, and this position should be maintained during the forced expiratory procedures; the patient should not
FVC/FEV1 ratio | pre the intervention and immediately after the intervention
  we recorded (FEV1) and (FVC) then we calculated the ratio between them
maximum voluntary ventilation (MVV) | pre the intervention and immediately after the intervention
  forced expiratory volume in the first second (FEV1) The patients were taught the following procedure of doing Pulmonary Function Test: 1) A clean mouthpiece was given to the patient and is attached to the valve at the end of the spirometer tubing. (2) The patient was wearing a nasal clip, sitting comfortably with his or her feet flat on the ground; (3) The proper chin neck posture was demonstrated to the patient: the chin should be lifted and the neck slightly extended, and this position should be maintained during the forced expiratory procedures
peak expiratory flow (PEF) in liter/min | pre the intervention and immediately after the intervention
  peak expiratory flow (PEF) The patients were taught the following procedure of doing Pulmonary Function Test: 1) A clean mouthpiece was given to the patient and is attached to the valve at the end of the spirometer tubing.. 2) The patient was wearing a nasal clip, sitting comfortably with his or her feet flat on the ground; (3) The proper chin neck posture was demonstrated to the patient: the chin should be lifted and the neck slightly extended, and this position should be maintained during the forced expiratory procedures;

OTHER OUTCOMES:
Arabic Oswestery Disability Index (AODI) for functional assessment | pre the intervention and immediately after the intervention
  Patients filled out a questionnaire that provides a percentage score of how well they functioned in everyday activities before and after sessions. This survey evaluates daily function in ten activities of daily living. The categories were scored from zero to five (6 categories). If all 10 sectors were finished the result is calculated as follows: if 20 the total result out of 50 total possible score x 100 = 40%.
  Scores: 1- Zero to twenty percent: Minimal disability. 2- Twenty one to forty percent: Moderate disability. 3- Forty one to sixty percent: Severe disability. 4- Sixty one to eighty percent: Crippled 5- Eighty one to one
weight | pre the intervention only
  we use weighing scale to measure weight of the subject in kilograms
age | pre the intervention only
  document the patient age through personal history information
height | pre the intervention only
  we measure height in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Delta University For Science and Technology, Al Manşūrah, Gamasah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided